CLINICAL TRIAL: NCT04683822
Title: Investigation of the Effectiveness of a Home Exercise Program Combined With Telerehabilitation in Pulmonary Hypertension Patients
Brief Title: Telerehabilitation in Patients With Pulmonary Hypertension
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Marmara University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 1443
Record Dates: First submitted 2020-12-20; First posted 2020-12-24 (Actual); Last update posted 2020-12-24 (Actual); Status verified 2020-12

CONDITIONS: Pulmonary Hypertension
MeSH Terms: conditions — Hypertension, Pulmonary | interventions — Telerehabilitation

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Exercise group (Experimental): Patients who receive telerehabilitaton
  Interventions: Other: Telerehabilitation
- Control (No Intervention): Patients with routine care

INTERVENTIONS:
Other: Telerehabilitation — Patients will attend telerehabilitation sessions
  Arms: Exercise group

SUMMARY:
Patients with pulmonary hypertension will be randomized into two groups. One group will receive telerehabilitation sessions including upper and lower extremity strengthening exercises and breathing exercises. The other will me monitored routinely. Patients will be assessed by 6 minute walk test, emphasis-10 questionnaire for quality of life and muscle strength with hand-held dynamometer.

ELIGIBILITY:
Inclusion Criteria:

* Patients with pulmonary hypertension

Exclusion Criteria:

* Patients with severe exercise intolerance
* Patients with musculoskeletal problems that hinder exercise
* Patients who refuse to join the study

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2021-01 (Estimated); Primary Completion 2021-05 (Estimated); Study Completion 2021-06 (Estimated)

PRIMARY OUTCOMES:
Muscle strength | 3 months
  Muscle strength measured with hand held dynamometer

IPD SHARING:
Plan to Share IPD: Undecided